CLINICAL TRIAL: NCT07104500
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, 78-Week Efficacy and Safety Study of VK2735 Administered Subcutaneously for Weight Management in Participants Without Type 2 Diabetes Who Are Obese, or Overweight With at Least One Weight-related Comorbid Condition
Brief Title: VK2735 for Weight Management Phase 3
Acronym: VANQUISH 1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Viking Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VK2735-301
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo Assignment (Placebo Comparator): VK2735 Placebo Comparator Once Weekly
  Interventions: Drug: VK2735
- Active Assignment (Dose 1) (Experimental): VK2735 7.5mg Once Weekly
  Interventions: Drug: VK2735
- Active Assignment (Dose 2) (Experimental): VK2735 12.5mg Once Weekly
  Interventions: Drug: VK2735
- Active Assignment (Dose 3) (Experimental): VK2735 17.5mg Once Weekly
  Interventions: Drug: VK2735

INTERVENTIONS:
Drug: VK2735 — VK2735 is a peptide GLP-1 and GIP dual agonist administered Once Weekly

SUMMARY:
This is a phase 3, multicenter, 78-week randomized, double-blind, placebo-controlled, parallel arm study that will evaluate the weight loss efficacy as well as safety, tolerability, pharmacodynamic effects, and pharmacokinetics of VK2735 in adults who are obese (BMI ≥30 kg/m2) or overweight (BMI ≥27 kg/m2) with one or more weight related comorbid condition without Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age at the time of signing the informed consent
2. Body mass index (BMI) ≥30 kg/m2 OR ≥27 kg/m2 with at least one weight-related co- morbid condition (treated or untreated)

   * Weight-related co-morbid conditions include hypertension, dyslipidemia, obstructive sleep apnea or cardiovascular disease
   * Cardiovascular disease includes, for example, ischemic cardiovascular disease, New York Heart Association (NYHA) Functional Class I-III heart failure
   * BMI calculated at the Screening visit will be used to determine eligibility

Exclusion Criteria:

1. History of or current clinically significant medical disorder that, in the opinion of the Investigator, does not support study participation
2. Self-reported body weight change of 5% or more within 3 months of screening
3. Have a prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty if performed >1 year prior to screening)
4. Have or plan to have endoscopic and/or device-based therapy for obesity or have had device removal within the last 6 months prior to screening (such as, mucosa ablation, gastric artery embolization, intragastric balloon, duodenal-jejunal endoluminal line)
5. Current or past diagnosis of diabetes mellitus (including type 1, type 2, except gestational diabetes)
6. Treatment with glucose-lowering agent(s) within 90 days before screening
7. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2)
8. History of acute or chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline for participants receiving VK2735 after 78 weeks of treatment | 78 Weeks

SECONDARY OUTCOMES:
Percentage of participants who achieve ≥5%, ≥10%, ≥15% and ≥20% body weight reduction after 78 weeks of treatment | 78 Weeks

CONTACTS AND LOCATIONS:
Locations (137):
- United States (135):
  - Viking Clinical Site #1037, Birmingham, Alabama
  - Viking Clinical Site #1064, Birmingham, Alabama
  - Viking Clinical Site #1128, Huntsville, Alabama
  - Viking Clinical Site #1081, Mobile, Alabama
  - Viking Clinical Site #1005, Chandler, Arizona
  - Viking Clinical Site #1017, Flagstaff, Arizona
  - Viking Clinical Site #1018, Peoria, Arizona
  - Viking Clinical Site #1135, Scottsdale, Arizona
  - Viking Clinical Site #1019, Tucson, Arizona
  - Viking Clinical Site #1036, Little Rock, Arkansas
  - Viking Clinical Site #1071, Chula Vista, California
  - Viking Clinical Site #1070, Escondido, California
  - Viking Clinical Site #1054, Huntington Park, California
  - Viking Clinical Site #1014, Lake Forest, California
  - Viking Clinical Site #1129, Lemon Grove, California
  - Viking Clinical Site #1051, Lincoln, California
  - Viking Clinical Site #1050, Long Beach, California
  - Viking Clinical Site #1055, Los Angeles, California
  - Viking Clinical Site #1078, Manteca, California
  - Viking Clinical Site #1053, Montclair, California
  - Viking Clinical Site #1068, Panorama City, California
  - Viking Clinical Site #1132, Rolling Hills Estates, California
  - Viking Clinical Site #1131, San Diego, California
  - Viking Clinical Site #1104, Santa Maria, California
  - Viking Clinical Site #1052, Spring Valley, California
  - Viking Clinical Site #1109, Tustin, California
  - Viking Clinical Site #1067, Van Nuys, California
  - Viking Clinical Site #1079, Walnut Creek, California
  - Viking Clinical Site #1119, Denver, Colorado
  - Viking Clinical Site #1123, Washington D.C., District of Columbia
  - Viking Clinical Site #1013, Clearwater, Florida
  - Viking Clinical Site #1121, Clearwater, Florida
  - Viking Clinical Site #1003, Cooper City, Florida
  - Viking Clinical Site #1112, DeLand, Florida
  - Viking Clinical Site #1107, Delray Beach, Florida
  - Viking Clinical Site #1083, Fort Myers, Florida
  - Viking Clinical Site #1058, Jacksonville, Florida
  - Viking Clinical Site #1076, Lakeland, Florida
  - Viking Clinical Site #1060, Lakewood Rch, Florida
  - Viking Clinical Site #1117, Miami, Florida
  - Viking Clinical Site #1059, New Port Richey, Florida
  - Viking Clinical Site #1012, Ocoee, Florida
  - Viking Clinical Site #1056, Palmetto Bay, Florida
  - Viking Clinical Site #1011, Port Orange, Florida
  - Viking Clinical Site #1057, West Palm Beach, Florida
  - Viking Clinical Site #1116, Atlanta, Georgia
  - Viking Clinical Site #1030, Columbus, Georgia
  - Viking Clinical Site #1120, Rincon, Georgia
  - Viking Clinical Site #1093, Savannah, Georgia
  - Viking Clinical Site #1025, Woodstock, Georgia
  - Viking Clinical Site #1062, Honolulu, Hawaii
  - Viking Clinical Site #1080, Meridian, Idaho
  - Viking Clinical Site #1006, Chicago, Illinois
  - Viking Clinical Site #1090, Chicago, Illinois
  - Viking Clinical Site #1138, Westmont, Illinois
  - Viking Clinical Site #1127, Valparaiso, Indiana
  - Viking Clinical Site #1022, West Des Moines, Iowa
  - Viking Clinical Site #1099, Wichita, Kansas
  - Viking Clinical Site #1069, Lexington, Kentucky
  - Viking Clinical Site #1040, Lexington, Kentucky
  - Viking Clinical Site #1009, Louisville, Kentucky
  - Viking Clinical Site #1118, Baton Rouge, Louisiana
  - Viking Clinical Site #1139, Baton Rouge, Louisiana
  - Viking Clinical Site #1106, Lafayette, Louisiana
  - Viking Clinical Site #1020, Metairie, Louisiana
  - Viking Clinical Site #1087, Monroe, Louisiana
  - Viking Clinical Site #1094, Chevy Chase, Maryland
  - Viking Clinical Site #1066, Rockville, Maryland
  - Viking Clinical Site #1103, Boston, Massachusetts
  - Viking Clinical Site #1001, Methuen, Massachusetts
  - Viking Clinical Site #1136, Needham, Massachusetts
  - Viking Clinical Site #1038, Ypsilanti, Michigan
  - Viking Clinical Site #1140, Gulfport, Mississippi
  - Viking Clinical Site #1031, City of Saint Peters, Missouri
  - Viking Clinical Site #1016, Kansas City, Missouri
  - Viking Clinical Site #1125, Springfield, Missouri
  - Viking Clinical Site #1108, St Louis, Missouri
  - Viking Clinical Site #1010, Butte, Montana
  - Viking Clinical Site #1075, Omaha, Nebraska
  - Viking Clinical Site #1035, Las Vegas, Nevada
  - Viking Clinical Site #1034, Reno, Nevada
  - Viking Clinical Site #1065, Lebanon, New Hampshire
  - Viking Clinical Site #1095, Marlton, New Jersey
  - Viking Clinical Site #1029, Albuquerque, New Mexico
  - Viking Clinical Site #1088, Albany, New York
  - Viking Clinical Site #1042, East Syracuse, New York
  - Viking Clinical Site #1096, Hartsdale, New York
  - Viking Clinical Site #1133, New York, New York
  - Viking Clinical Site #1142, New York, New York
  - Viking Clinical Site #1021, The Bronx, New York
  - Viking Clinical Site #1032, Westfield, New York
  - Viking Clinical Site #1141, Charlotte, North Carolina
  - Viking Clinical Site #1122, Durham, North Carolina
  - Viking Clinical Site #1144, Fayetteville, North Carolina
  - Viking Clinical Site #1026, Greensboro, North Carolina
  - Viking Clinical Site #1110, Morehead City, North Carolina
  - Viking Clinical Site #1061, Morehead City, North Carolina
  - Viking Clinical Site #1027, Fargo, North Dakota
  - Viking Clinical Site #1043, Cincinnati, Ohio
  - Viking Clinical Site #1074, Cincinnati, Ohio
  - Viking Clinical Site #1044, Cleveland, Ohio
  - Viking Clinical Site #1089, Columbus, Ohio
  - Viking Clinical Site #1113, Norman, Oklahoma
  - Viking Clinical Site #1137, Tulsa, Oklahoma
  - Viking Clinical Site #1102, Medford, Oregon
  - Viking Clinical Site #1097, Portland, Oregon
  - Viking Clinical Site #1126, Portland, Oregon
  - Viking Clinical Site #1045, East Greenwich, Rhode Island
  - Viking Clinical Site #1028, Greenville, South Carolina
  - Viking Clinical Site #1134, Myrtle Beach, South Carolina
  - Viking Clinical Site #1023, North Charleston, South Carolina
  - Viking Clinical Site #1004, Knoxville, Tennessee
  - Viking Clinical Site #1008, Nashville, Tennessee
  - Viking Clinical Site #1047, Abilene, Texas
  - Viking Clinical Site #1063, Austin, Texas
  - Viking Clinical Site #1007, Austin, Texas
  - Viking Clinical Site #1091, Bellaire, Texas
  - Viking Clinical Site #1124, Brownsville, Texas
  - Viking Clinical Site #1049, Dallas, Texas
  - Viking Clinical Site #1048, Dallas, Texas
  - Viking Clinical Site #1111, Frisco, Texas
  - Viking Clinical Site #1046, Houston, Texas
  - Viking Clinical Site #1077, Lampasas, Texas
  - Viking Clinical Site #1143, San Antonio, Texas
  - Viking Clinical Site #1085, San Antonio, Texas
  - Viking Clinical Site #1073, San Antonio, Texas
  - Viking Clinical Site #1101, Waco, Texas
  - Viking Clinical Site #1002, Ogden, Utah
  - Viking Clinical Site #1092, Salt Lake City, Utah
  - Viking Clinical Site #1039, Sandy City, Utah
  - Viking Clinical Site #1024, St. George, Utah
  - Viking Clinical Site #1098, Arlington, Virginia
  - Viking Clinical Site #1082, Suffolk, Virginia
  - Viking Clinical Site #1072, Renton, Washington
  - Viking Clinical Site #1041, Spokane, Washington
- Puerto Rico (2):
  - Viking Clinical Site #1130, Mayagüez
  - Viking Clinical Site #1086, San Juan